CLINICAL TRIAL: NCT00392275
Title: Penetrance of Third Generation Fluoroquinolones in Eyes With Functioning Filtering Blebs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0208-29
Record Dates: First submitted 2006-10-23; First posted 2006-10-25 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2007-12

CONDITIONS: Cataract
Keywords: Cataract; Aqueous absorption; Funtioning Filtering Blebs
MeSH Terms: conditions — Cataract | interventions — Ofloxacin; Ciprofloxacin; Levofloxacin

INTERVENTIONS:
Drug: Ofloxacin 0.3%
Drug: Ciprofloxacin 0.3%
Drug: Levofloxacin 0.5%
Drug: Ofloxacin 400mg
Drug: Ciprofloxacin 400mg
Drug: Levofloxacin 250mg

SUMMARY:
Based on previous results with eyes without filtering blebs, the aqueous concentrations of ofloxacin and levofloxacin will exceed the concentration of ciprofloxacin after either topical or topical plus oral administration.

DETAILED DESCRIPTION:
The purpose of this study is to assay human aqueous for concentrations of ofloxacin, ciprofloxacin and levofloxacin after topical or combined topical and oral administration in eyes with filtering blebs.

ELIGIBILITY:
Inclusion Criteria:

* All patients with functioning filtering blebs will be evaluated prospectively for inclusion

Exclusion Criteria:

* Any subject who is already scheduled to have cataract surgery performed will qualify for participation with the exception of the following exclusion criteria:

  * Ongoing ocular inflammatory disease
  * Bleb leakage - determined by Seidel test
  * Suspected infection
  * Known contraindications to use of any of these study medications.
  * Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48
Dates: Start 2002-11; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Aqueous levels of antibiotics

CONTACTS AND LOCATIONS:
Overall Officials: Louis B Cantor, MD, Principal Investigator — Indiana University
Locations (3):
- United States (3):
  - Indiana University Hospital, Indianapolis, Indiana
  - Richard L Rodeboush VA Medical Center, Indianapolis, Indiana
  - Wishard Memorial Hospital, Indianapolis, Indiana

REFERENCES:
- [Background] Cantor LB, Donnenfeld E, Katz LJ, Gee WL, Finley CD, Lakhani VK, Hoop J, Flarty K. Penetration of ofloxacin and ciprofloxacin into the aqueous humor of eyes with functioning filtering blebs: a randomized trial. Arch Ophthalmol. 2001 Sep;119(9):1254-7. doi: 10.1001/archopht.119.9.1254. PMID 11545629
- [Derived] Cantor LB, WuDunn D, Yung CW, Valluri S, Catoira YP, Hoop JS, Morgan LS. Ocular penetration of levofloxacin, ofloxacin and ciprofloxacin in eyes with functioning filtering blebs: investigator masked, randomised clinical trial. Br J Ophthalmol. 2008 Mar;92(3):345-7. doi: 10.1136/bjo.2007.121541. Epub 2008 Jan 22. PMID 18211932